CLINICAL TRIAL: NCT01233180
Title: Randomized Controlled Trial Comparing Gua Sha Massage and Thermotherapy for Chronic Neck Pain: Effects on Pain Intensity, Haptic Perception and Body Image.
Brief Title: Effects of Gua Sha and Thermotherapy on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Gustav J Dobos, MD, University of Duisburg-Essen, Chair of Complementary and Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-4434
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Neck Pain
Keywords: neck pain; massage; hyperthermia, induced; touch perception; randomized controlled trial
MeSH Terms: conditions — Neck Pain; Hyperthermia | interventions — Hyperthermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gua Sha (Active Comparator): Single Gua Sha treatment of the neck and shoulder region.
  Interventions: Other: Gua Sha
- Thermotherapy (Active Comparator): Single use of a mud heat pad on the neck and shoulder region.
  Interventions: Device: Thermotherapy

INTERVENTIONS:
Other: Gua Sha — Single Gua Sha treatment of the neck and shoulder region
  Arms: Gua Sha
Device: Thermotherapy — Single use of a mud heat pad on the neck and shoulder region
  Arms: Thermotherapy

SUMMARY:
Gua Sha massage is a traditional chinese medical treatment. It is mostly used in the treatment of the common cold and pain syndromes. Gua Sha involves pressuring the skin by a round-edged instrument until small petechiae appear. This so called "sha", considered as the removal of blood stasis by traditional practitioners, will fade within a few days. Normally, this treatment is not considered as painful, but as relaxing and easing tense muscles.

In this study, the investigators will investigate the effectivity of Gua Sha massage in treating chronic neck pain. The investigators will research effects on subjective pain intensity, neck pain specific disability and haptic perception.

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical neck pain, at least 40 mm on a 100mm visual analog scale.
* Pain for at least 3 months.

Exclusion Criteria:

* radicular symptoms
* congenital spine deformity
* pregnancy
* rheumatic diseases
* oncologic diseases
* other severe psychiatric or somatic comorbidity
* recent invasive or surgical treatment of the spine
* participation in other studies
* skin diseases in the area to be treated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity (100mm visual analog scale) | Day 4

SECONDARY OUTCOMES:
Neck disability index (NDI) | Day 4
  The Neck Disability Index is an instrument to assess neck pain complaints.
  Reference: Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther 1991;14:409-415.
Haptic perception | Day 4
  The design consists of two angle legs, of which one angle leg has to be readjusted to a given angle adjustment. This is done by haptic perception without visual feedback. The deviation of the adjusted angle from the locked angle is measured.
  Reference: Grunwald, M., Ettich, C., Busse, F., Assmann, B., Dähne, A., Gertz, H.-J., (2002): Angle paradigm: A new method to measure right parietal dysfunctions in anorexia nervosa. Archives of Clinical Neuropsychology , 17, pp. 485- 496

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Knappschafts-Krankenhaus, Department for Internal and Integrative Medicine, Essen, North Rhine-Westphalia, Germany